CLINICAL TRIAL: NCT06540391
Title: A Phase 1b, Randomized, Open-Label Trial to Evaluate Safety, Engraftment, and Initial Signs of Clinical Activity of MB097 in Combination With Pembrolizumab in Melanoma Patients With Primary Resistance to an AntiPD1Containing Immunotherapy
Brief Title: A Phase 1b Trial to Evaluate Safety of MB097 in Combination With Pembrolizumab in Melanoma Patients
Acronym: MELODY-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Microbiotica Ltd (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB097-01; KEYNOTE-E75 (Other: Merck Sharp & Dohme LLC); MK-3475-E75 (Other: Merck Sharp & Dohme LLC); 2023-507377-17 (EudraCT Number)
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Vancomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MB097 and pembrolizumab (Experimental): MB097 PO (2 capsules once a day) for 6 months Pembrolizumab IV 200mg Q3W for 6 months
  Interventions: Biological: MB097; Biological: Pembrolizumab
- MB097 and pembrolizumab with vancomycin preconditioning (Experimental): Vancomycin 125mg QID for 5 days plus 2 day wash-out prior to receiving MB097 PO (2 capsules once a day) for 6 months Pembrolizumab IV 200mg Q3W for 6 months
  Interventions: Biological: MB097; Biological: Pembrolizumab; Drug: Vancomycin
- Extended treatment (Experimental): Patients experiencing clinical benefit may continue to receive study intervention (pembrolizumab only IV 200mg Q3W) until such time as a criterion for discontinuation is met or 35 doses of pembrolizumab have been administered.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: MB097 — Live bacterial therapeutic for oral administration
  Arms: MB097 and pembrolizumab; MB097 and pembrolizumab with vancomycin preconditioning
Biological: Pembrolizumab — IV infusion
  Other Names: KEYTRUDA®
Drug: Vancomycin — Antibiotic
  Arms: MB097 and pembrolizumab with vancomycin preconditioning

SUMMARY:
A Phase 1b study to evaluate the safety and tolerability of MB097 given in combination with pembrolizumab in patients with melanoma who demonstrate primary resistance to anti-PD1 therapy.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Must have primary resistant cutaneous melanoma and have experienced disease progression as defined by RECIST v1.1 after receiving at least 6 weeks of exposure to PD-1/PD-L1 inhibitor therapy, generally correlating with 2 complete cycles of PD-1/PD-L1 inhibitor therapy.
* Must have histological or cytological confirmation of Stage III (unresectable) or Stage IV cutaneous melanoma
* Must have radiographically measurable disease per RECIST v1.1
* Must be at least 18 years of age at time of informed consent
* Must provide written informed consent, according to local guidelines, signed and dated by the patient prior to the performance of any study-specific procedures, sampling, or analysis
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 at time of informed consent.
* Must have acceptable organ function, as evidenced by laboratory data prior to first dose of any study drug
* Female patients must not be lactating or pregnant
* Male patients, and female patients of childbearing potential who are at risk of pregnancy must agree to use a highly effective method of contraception
* Must have life expectancy ≥12 weeks after the start of any study drug per Investigator's judgment
* Must be willing and able to comply with the Protocol, scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines, and all other study procedures.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following

* Any treatment for melanoma following the failure of an aPD-1-containing treatment, i.e., no intervening treatments between aPD-1 failure and enrollment into study;
* Prior therapy with any of the following:

  * Radiation therapy to target lesions within 6 weeks of the first dose of MB097
  * Major invasive surgery, excluding placement of vascular access, within 28 days of the first dose of any study drug
  * Probiotic supplement use within 7 days of the first dose of any study
  * LBP use, including FMT, within 6 months of start of therapy with MB097.
* Active, uncontrolled infection requiring systemic antimicrobial, antiviral, or antifungal therapy.
* Active, uncontrolled, symptomatic brain metastases or leptomeningeal metastases
* Ocular, uveal, acral, or mucosal melanoma
* Prior treatment-related toxicities that have not resolved to Grade 2 or less per NCI CTCAE v5.0;
* Patients with a history of immune-related colitis may be included if symptoms have resolved to Grade 1 or less for at least 14 days prior to screening
* Any history of CTCAE v5.0 immune-related toxicity Grade 3 or greater from prior CPI that is recurrent or steroid-refractory
* Known hypersensitivity to any of the ingredients of the study drug(s) or known hypersensitivity to vancomycin (oral or IV)
* Significant medical conditions which, in the Investigator's opinion, could compromise or interfere with the patient's safety or integrity of the study outcomes
* Severe colitis of any etiology (except colitis associated with treatment with an aPD-1 inhibitor)
* History of another malignancy within 3 years before the first dose of any study drug, or any evidence of residual disease from a previously diagnosed malignancy
* Clinically significant (i.e., active) cardiovascular disease
* Any clinically significant safety concern related to prior CPI therapy
* Active autoimmune disease that required systemic treatment in the past 2 years prior to screening
* History of investigational agent or device use within 4 weeks prior to the first dose of study treatment or current participation in a study of an investigational agent
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation, or, in the opinion of the Investigator, is considered to not be in the best interest of the patient to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of MB097 in combination with pembrolizumab | From Visit 1 to 30 days after the last dose of study treatment
  Assessed by the following:
  * The incidence and severity of treatment-emergent AEs (TEAEs) per NCI CTCAE v5.0;
  * Immune-related AEs (irAEs);
  * AESIs; and
  * Any clinically significant abnormalities in laboratory results, physical examination findings, 12-lead ECG findings, and vital signs using the NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Best objective response rate (b-ORR) by RECIST v1.1 and iRECIST | Up to Week 24 or Week 105(for patients in extended treatment)
  b-ORR is the best response recorded from the start of the treatment until disease progression/recurrence (Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD))
Overall response rate (ORR) by RECIST v1.1 and iRECIST | Up to Week 24 or Week 105(for patients in extended treatment)
  Overall response of CR, PR, SD or PD.
Disease control rate (DCR) by RECIST v1.1 and iRECIST | Up to Week 24 or Week 105(for patients in extended treatment)
  DCR is defined as the proportion of patients with CR, PR, or SD for 8 weeks or more, by RECIST v1.1 and iRECIST
Duration of response | Up to Week 24 or Week 105(for patients in extended treatment)
  The time from first objective response until progression of disease or death
Progression-free survival, | Up to Week 24 and Week 36, and Week 105(for patients in extended treatment)
  The time from enrollment until disease progression or death
Time to progression | Up to Week 24 or Week 105(for patients in extended treatment)
  Time until disease progression and overall survival
Quantification of MB097 strains at baseline and over the intervention period in patients treated with MB097 with and without vancomycin preconditioning and correlation to efficacy measures | Up to Week 24 or Week 105(for patients in extended treatment)

CONTACTS AND LOCATIONS:
Locations (19):
- France (5):
  - Centre Georges Francois Leclerc, Dijon
  - CHU de Lille - Hopital Claude Huriez, Lille
  - Centre Leon Berard, Lyon
  - AP-HM - Hopital de la Timone, Marseille
  - HCL Centre Hospitalier Lyon Sud, Pierre-Bénite
- Italy (3):
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Istituto Clinico Humanitas, Rozzano
- Spain (4):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - South Texas Accelerated Research Therapeutics (START) Madrid - CIOCC, Madrid
  - Consorcio Hospital General Universitario de Valencia, Valencia
- United Kingdom (7):
  - Sussex Cancer Centre, Brighton
  - Addenbrooke's Hospital, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Freeman Hospital, Newcastle
  - Royal Marsden Hospital - Surrey, Sutton